CLINICAL TRIAL: NCT04846608
Title: Descriptive Study of Emergency Room Visits From Nursing Home Residents for Behavioral Problems at the Nancy University Hospital: Place of the Advanced Practice Nurse
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Marie MANGEOT- Nurse (Unknown); Mahmut GUNDESLI MD (Unknown)
Responsible Party: Principal Investigator, Bernadette HANESSE, MD, Central Hospital, Nancy, France
Other Study IDs: 2021PI027
Record Dates: First submitted 2021-03-26; First posted 2021-04-15 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Behavioral Disorders
MeSH Terms: conditions — Mental Disorders | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nursing home residents with behavioural problems: Nursing home residents from Grand Nancy aged 75 and over referred to emergency departments for disorientation, agitation, dementia or behavioural problems during the study period
  Interventions: Other: Observation
- Nursing home residents with other problems: Nursing home residents from Grand Nancy aged 75 and over referred to emergency departments for other reasons
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observation

SUMMARY:
The demographic evolution of old age is a reality. After the age of 75, 2 out of 3 people living in institutions have neurocognitive disorders. Behavioural disorders such as physical aggression, agitation, hallucinations, sleep disorders, generate difficulties in the management of these patients and lead to unscheduled emergency hospitalizations. Non-pharmacological management of behavioral disorders is recommended as a first-line treatment because of its low risk and potential improvement (Haute Autorité de Santé 2009). However, this management is not simple and obvious to put in place, especially since not all elderly people with Behavioural disorders are in adapted structures. The advanced practice nurse specializing in geriatrics has a place in this care pathway. Because of her skills, she could "organize multi-professional care, set up analyses of practices within the nursing homes, train caregivers appropriately, and limit hospitalizations due to behavioral problems" (SALIEGE L. 2020). Advanced practice nursing is in its infancy in France, and everything remains to be done (International Council of Nurses- directive). The aim of the study is to identify the number of emergency room visits by people aged 75 and over for behavioral problems in nursing home during a 6 month-period.

ELIGIBILITY:
Inclusion Criteria:

* Person who has received full information on the organization of the research and has not objected to the use of this data
* Elderly men and women 75 years of age and older at the time of the emergency room visit
* Having for main residence one of the nursing homes of the Grand Nancy
* Administratively present in the emergency department
* Having been admitted to the emergency room for the following reasons:

  * Behavioural problems
  * Agitation
  * Dementia
  * Disorientation
  * Delirium

Exclusion Criteria:

* People under 75 years of age
* Residing at home or in a senior residence or in a nursing home outside Grand Nancy
* Referred by an inpatient department (rehabilitation department)
* Other reasons for emergency room use such as "depression" and "apathy

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All persons aged 75 and over, residents of nursing homes in the Nancy area, who consulted the emergency department during the 6 month study period
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Number of passage of people aged 75 and over referred to emergency departments by nursing homes for disorientation, agitation, dementia or behavioural problems during the study period | through study completion, an average of 6 months
  Number of passage of people aged 75 and over referred to emergency departments by nursing homes for disorientation, agitation, dementia or behavioural problems during the study period

SECONDARY OUTCOMES:
Age of the patients | through study completion, an average of 6 months
Gender of the patients | through study completion, an average of 6 months
Presence of previous medical cognitive disorder | through study completion, an average of 6 months
Name of nursing home of origin | through study completion, an average of 6 months
Length of stay at emergency room | through study completion, an average of 6 months
Referral after visit at emergency room | through study completion, an average of 6 months
Number of iterative passage of people aged 75 and over referred to emergency departments by nursing homes for disorientation, agitation, dementia or behavioural problems during the study period | through study completion, an average of 6 months
Presence of intervention of geriatric mobile team | through study completion, an average of 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de NANCY, Nancy, France

IPD SHARING:
Plan to Share IPD: No